CLINICAL TRIAL: NCT03493620
Title: Multicenter Randomized Prospective Study With Sham Group to Evaluate the Efficacy and Results of Endoscopic Gastroplasty Using Overstitch in Patients With Class I and II Obesity
Brief Title: Efficacy and Results of Endoscopic Gastroplasty Using Overstitch in Patients With Class I and II Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ApolloSham
Record Dates: First submitted 2018-03-14; First posted 2018-04-10 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device arm (Experimental): Gastric endosuturing will be performed until the entire gastric body is sutured in the form of a tube.
  Interventions: Procedure: Device arm
- Sham arm (Sham Comparator): Group II is a control group (only the endoscopist will know which group each patient belongs to)
  Interventions: Procedure: Sham arm

INTERVENTIONS:
Procedure: Device arm — Make a gastric tube (endoscopic sleeve gastroplasty) using the Apollo Overstitch suturing device through endoscopy.
  Arms: Device arm
Procedure: Sham arm — Group II will be conducted identically to Group I except for the procedure itself, and only the endoscopist, that is the researcher, will be aware of which group each patient belongs to.
  Arms: Sham arm

SUMMARY:
Obesity is a chronic disease that has grown to epidemic proportions in Brazil and throughout the world in recent years. Bariatric surgery has been the most effective method for the treatment and prophylaxis of complications caused by morbid obesity, thereby increasing the longevity and quality of life of patients. The treatment of patients with Class III obesity or higher or Class II with comorbidities is already well established with bariatric surgery being the best option. However, there is no consensus as to the best treatment in cases of Class I or II obesity without comorbidities. The objective of this research will be to make a gastric tube similar to that obtained by surgical gastroplication but using endoscopic intragastric sutures.

DETAILED DESCRIPTION:
The primary objective of this research will be to make a gastric tube similar to that obtained by surgical gastroplication but using endoscopic intragastric sutures. The secondary objective will be to correlate demographic, endoscopic and laboratory data with the outcomes.

This study will be carried out in two institutions. The Kaiser Clinic and Day Hospital and the Faculty of Medicine of ABC. Sixty patients will be randomly selected for treatment by Endospore Endoscopy (ESG) or as controls (only the endoscopist will know which group each patient belongs to). The draw will take place only after upper endoscopy has been carried out to avoid possible contraindications for the procedure due to injuries. Once the criteria for endoscopic evaluation have been met, randomization will be carried out in loco with the patient still sedated. Gastric Endo Sutures will be performed when the patient is randomized for Group I; Group II will be the control group. All patients will be followed up for two years by a multidisciplinary team (endoscopist, surgeon, nutritionist and psychologist). The data will be obtained during the outpatient follow-up at the Hospital Mario Covas and will include demographic (gender, age), clinical (height, weight, BMI, time after procedure, hypertension, diabetes, dyslipidemia, smoking, alcoholism) and operative data (complications).

Preparation to perform the examination/procedure: All exams will be performed with the patients within eight hours. The procedure will begin with the patient in left lateral decubitus position and under general anesthesia performed by an anesthesiologist. Endoscopic suturing will be performed with 2-0 prolene stitches until a tubular-shaped stomach is formed similar to vertical gastrectomy.

Recovery after the procedure: After this procedure and recovery from the anesthesia, all patients will only be discharged in the company of a companion. All patients will be counseled to enter in touch with the physician to report any signs or symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years,
* BMI > 30 and < 36 kg/m2, with or without comorbidities,
* BMI > 36 and < 40 without comorbidities

Exclusion Criteria:

* Previous gastric surgery
* Taking anticoagulant drugs
* Psychiatric disorders
* Severe esophagitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | outcome will be evaluated for 2 years
  weight in kg

SECONDARY OUTCOMES:
Weight maintenance | 2 years
  weight in kg
Surgical related complications | 2 years
Comorbidities | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Gustavo de Quadros, MD, Principal Investigator — Kaiser Clinica and Day Hospital; Eduardo Grecco, MD, Principal Investigator — ABC Medical School; Manoel Galvao Neto, MD, Principal Investigator — ABC Medical School; Thiago Ferreira de Souza, PhD, Principal Investigator — ABC Medical School
Locations (2):
- Brazil (2):
  - Faculty of Medicine of ABC, Santo André, São Paulo
  - Kaiser Clinic and Day Hospital, São José do Rio Preto, São Paulo